CLINICAL TRIAL: NCT04485338
Title: Radiographic Assessment of Lung Edema in Invasively Ventilated COVID-19 Patients (RALE-COVID) - Protocol for an International Multicenter Retrospective Study
Brief Title: Chest Radiography in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: University of Bari Aldo Moro (Other); Mahidol University (Other); Universitair Ziekenhuis Brussel (Other); Chonburi hospital (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. M.J. Schultz, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: RALE-COVID
Record Dates: First submitted 2020-07-23; First posted 2020-07-24 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Covid19
Keywords: Chest radiography; RALEscore; Radiographic Assessment of Lung Edema; ICU; invasively ventilated
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the prognostic performance of the RALE score with respect to duration of ventilation, and to describe changes in the RALE score over time.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an ICU participating in this study between December 1, 2019 and May 31, 2020
* Having had received invasive ventilation
* Having had received at least one chest radiograph under invasive ventilation
* Confirmed novel coronavirus diseases (COVID-19)

Exclusion Criteria:

- Age < 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Severe COVID-19 patients under invasive ventilation who received as part of standard care and routine imaging.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
The prognostic capacity of the Radiographic Assessment of Lung Edema (RALE) score of the first CXR under invasive ventilation in patients with severe COVID-19. | 90 days

SECONDARY OUTCOMES:
The prognostic capacity of changes in the RALE score of consecutive CXRs under invasive ventilation in patients with severe COVID-19 | 90 days
Number of ventilator-free day and alive at day 28 (VFD) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J. Schultz, Prof., Principal Investigator — Amsterdam University Medical Centers, location 'AMC'
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided